CLINICAL TRIAL: NCT01245660
Title: Pilot Study of Lapatinib (Tyverb®) in Neoadjuvant Treatment for Patients With Locally Bladder Carcinoma Before Cystectomy
Brief Title: A Phase 0 of Neoadjuvant Lapatinib in Infiltrative Bladder Carcinoma Before Cystectomy
Acronym: LAPAINBLAD
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: The rythm of enrollment was not compatible with the objective of recruitement in the research.
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: CHUBX 2009/04
Record Dates: First submitted 2010-11-18; First posted 2010-11-22 (Estimated); Last update posted 2013-01-11 (Estimated); Status verified 2013-01

CONDITIONS: Bladder Carcinoma; Infiltrative Bladder Carcinoma; Cystectomy
Keywords: Phase 0; Bladder carcinoma; egf pathway; infiltrative bladder carcinoma; cystectomy; LAPATINIB
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Lapatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Patient (Experimental)
  Interventions: Drug: LAPATINIB

INTERVENTIONS:
Drug: LAPATINIB — Lapatinib, 1250 mg per day, per os, during 3 weeks +/- 5 days.

SUMMARY:
Modification of the EGF signalling pathway and / or HER 2, by Lapatinib in bladder cancer.

DETAILED DESCRIPTION:
Patients with invasive bladder tumor , candidates for radical cystectomy. Patients will receive Lapatinib during 3 weeks +/- 5 days, before cystectomy. A comparison of tissue from the original biopsy and cystectomy after Lapatinib will allow this to occur.

TREATMENT AND STRATEGY Lapatinib in bladder carcinoma -Overall there are arguments for considering that egf pathway is involved in bladder carcinoma and so far that drugs inhibiting EGF pathway could have an impact for therapeutical endpoints.

Nevertheless it is unclear that from previous studies that adding egf inhibiting drug to chemotherapy is clinically relevant, essentially by difficulties to measure a beneficial endpoint while downstream EGF pathways have been modified by these drugs, as shown with lapatinib (see 2.1.5).

Furthermore, there is no argument for initial selection of patients based on the initial egfr and/or her 2 tumor profile, asking for more intense knowledge.

LAPATINIB TREATMENT Patients will receive lapatinib therapy at a daily standard dose of 1500 mg.

LAPATINIB TREATMENT DURATION Patients will then receive 3 weeks of lapatinib therapy + possible 5 days. As the study is a non direct benefit study, the exposition to the drug is proposed during the standard window of 3 to 4 weeks to organize a radical cystectomy in patients with muscle invasive bladder carcinoma. In this study patients, the standard procedure is not delayed for the purpose of the study.

The duration of exposition to lapatinib as to be long enough to have a continuous impact of biological events to induce indeed inhibition of EGF pathway but also to impact on more complex or more distal events as apoptosis and so to be able to measure it. This justifies a 3 weeks of treatment + possible up to 5 days more due to surgical organization procedures.

Surgery will take place on the last day of treatment, which is recommended due to the half-life of lapatinib. Nevertheless for surgical purpose, the drug could be not given on the day of surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients must sign and date IRB/EC-approved informed consent,
* Age ≥ 18
* Patients must have a life expectancy of at least 6 months,
* Patients must have a Karnofsky performance status ≥ 80%,
* Clinical stage T2NxM0 to T4aNxM0 bladder cancer
* Muscle-invasive transitional cell carcinoma by histology (focal squamous and/or adenocarcinoma differentiation defined as ≤ 10% of tumor volume allowed, sarcomatoid and small-cell components not allowed)
* Considered to have a macroscopic residue in the bladder to allow comparison of tissue samples at cystectomy to initial biopsies
* Candidates for radical cystectomy
* Patient with normal cardiac function, LVEF ≥ 50% measured by echocardiography or MUGA scan
* Able to swallow and retain oral medication
* A female is eligible to enter and participate in this study if she is of : Non-child-bearing potential (i.e., a woman with functioning ovaries who have a current documented tubal ligation or hysterectomy or a woman who is menopausal), or Child-bearing potential (i.e. a woman with functioning ovaries and no documented impairment of oviductal or uterine function that would cause sterility. This category includes women with oligomenorrhoea (even severe), women who are perimenopausal and young women who have begun to menstruate), who have a negative serum pregnancy test at screening, and agree to one of the following consistent and correct use of one acceptable methods of birth control : Any intrauterine device (IUD) with a documented failure rate of less than 1% per year, or combined oral contraception
* care must be taken to avoid pregnancy in partners of male patients.
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures.
* Affiliated or profit patient of a social security system

Exclusion Criteria:

* Prior pelvic radiation or neoadjuvant chemotherapy.
* Pregnancy or breastfeeding.
* Other severe acute or chronic medical or psychiatric condition that would impart, in the judgment of the investigator, excess risk associated with study participation or study drug administration, or which, in the judgment of the investigator, would make the patient inappropriate for entry into this study.
* Patients with significantly reduced LVEF or LVEF < 50%.
* Patient with any of the following liver abnormal laboratory test :
* Serum bilirubin > 1,5 x upper limit of normal (ULN) (in case of Gilbert syndrome, a higher serum total bilirubin (< 2 ULN) is allowed
* Alanine amino transferase (ALAT) or aspartate amino transferase (ASAT) > 2,5 ULN
* Platelets <100 x 109/L, hemoglobin < 9 g/dl, absolute neutrophil count (ANC) <1.5 x 109/L
* Have current active hepatic or biliary disease (with exception of patients with Gilbert's syndrome, asymptomatic gallstones, liver metastases or stable chronic liver disease per investigator assessment)
* Serum creatinine > 1.5 x ULN.
* Previous therapy targeting EGFR or HER-2.
* Predominantly non transitional cell histology.
* Diagnosis of any second malignancy within the last 3 years, except basal cell carcinoma, squamous cell skin cancer, or in situ carcinoma of the cervix uteri that has been adequately treated with no evidence of recurrent disease for 12 months.
* Malabsorption syndrome, disease significantly affecting gastrointestinal function, or major resection of the stomach or bowel, that could affect absorption of lapatinib.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to lapatinib
* Uncontrolled inter-current illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, that would limit compliance with study requirements.
* History of uncontrolled or symptomatic angina
* History of arrhythmias requiring medications, or clinically significant, with the exception of asymptomatic atrial fibrillation requiring anticoagulation
* Myocardial infarction < 6 months from study entry
* Uncontrolled or symptomatic congestive heart failure
* Ejection fraction below the institutional normal limit
* Any other cardiac condition, which in the opinion of the treating physician, would make this protocol unreasonably hazardous for the patient
* Use of an investigational agent within 30 days or 5 half-lives, whichever is the longer, preceding the first dose of investigational product.
* Concurrent treatment with an investigational agent
* Concurrent treatment with cytotoxic chemotherapy, immunotherapy, biologic therapy, hormonal therapy or curative radiotherapy for locally advanced or metastatic TCC of the urothelial tract.
* Concomitant requirement for medication classified as CYP3A4 inducers or inhibitors.
* Patient under safeguard of justice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2011-01; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Effect on egf pathway at a molecular level of 3 weeks treatment by lapatinib. | At surgery (day 21-27)
  The primary objective of the study is to evaluate the effect at a molecular level, of 3 weeks of neoadjuvant lapatinib, in locally advanced muscle-invasive transitional cell carcinoma of the bladder. A comparison of tissue from the original biopsy and cystectomy after lapatinib will allow this to occur. This effect will be evaluated by studying proliferation and apoptotic markers as well as the phosphorylation of proteins which are components of the egf signalling pathway.

SECONDARY OUTCOMES:
Lapatinib biological response on key molecules of the egf pathway (EGFR, ERBB2, AKT ERK as well as their phosphorylation status.) | At screening (day -10 before inclusion) , surgery (day 21-27) and Follow up visit surgery (day 42-62)
  Because the availability of large scale data, the correlation between lapatinib biological response and the molecular alteration of other molecules beside those involved in the egf pathway will be explored. i.e. key molecules of the pathway will also be studied at the protein level (EGFR, ERBB2, AKT ERK) as well as their phosphorylation status.
Histological response | At surgery (day 21-27)
  To evaluate the histological response to lapatinib at the time of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Geneviève CHENE, Pr, Study Chair — USMR Bordeaux
Locations (1):
- CHU Bordeaux - Hôpital Saint André - Department of Medical Oncology, Bordeaux, France

REFERENCES:
- [Background] Rodel C, Weiss C, Sauer R. Trimodality treatment and selective organ preservation for bladder cancer. J Clin Oncol. 2006 Dec 10;24(35):5536-44. doi: 10.1200/JCO.2006.07.6729. PMID 17158539
- [Background] Jimenez RE, Hussain M, Bianco FJ Jr, Vaishampayan U, Tabazcka P, Sakr WA, Pontes JE, Wood DP Jr, Grignon DJ. Her-2/neu overexpression in muscle-invasive urothelial carcinoma of the bladder: prognostic significance and comparative analysis in primary and metastatic tumors. Clin Cancer Res. 2001 Aug;7(8):2440-7. PMID 11489824
- [Background] Advanced Bladder Cancer (ABC) Meta-analysis Collaboration. Neoadjuvant chemotherapy in invasive bladder cancer: update of a systematic review and meta-analysis of individual patient data advanced bladder cancer (ABC) meta-analysis collaboration. Eur Urol. 2005 Aug;48(2):202-5; discussion 205-6. doi: 10.1016/j.eururo.2005.04.006. Epub 2005 Apr 21. PMID 15939524